CLINICAL TRIAL: NCT06086418
Title: Effect of Perineural Dexamethasone on the Duration of Popliteal Nerve Block for Anesthesia After Pediatric Ankle Surgery
Brief Title: Perineural Dexamethasone on the Duration of Popliteal Nerve Block for Anesthesia After Pediatric Ankle Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13/2023
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2024-04

CONDITIONS: Ankle Disease; Ankle Injuries; Foot Injury; Foot Diseases
MeSH Terms: conditions — Ankle Injuries; Foot Injuries; Foot Diseases | interventions — Sodium Chloride; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- placebo (Placebo Comparator): 0.2% ropivacaine for popliteal nerve block
  Interventions: Drug: 0.9 % Sodium Chloride
- 0.1mg/kg Dexamethasone (Active Comparator): 0.1mg/kg dexamethasone added to 0.2% ropivacaine for popliteal nerve block
  Interventions: Drug: 0.1mg/kg Dexamethasone
- 0,05mg/kg dexamethasone (Active Comparator): 0.05mg/kg dexamethasone added to 0.2% ropivacaine for popliteal nerve block
  Interventions: Drug: 0.05mg/kg Dexamethasone

INTERVENTIONS:
Drug: 0.9 % Sodium Chloride — administration of 0.5ml/kg of 0,2% ropivacaine + 0.01ml/kg 0.9% sodium chloride for the popliteal nerve block
  Other Names: placebo
  Arms: placebo
Drug: 0.1mg/kg Dexamethasone — administration of 0.5ml/kg of 0.2% ropivacaine with 0.1mg/kg Dexamethasone for the popliteal nerve block
  Other Names: large dose
  Arms: 0.1mg/kg Dexamethasone
Drug: 0.05mg/kg Dexamethasone — administration of 0.5ml/kg of 0.2% ropivacaine with 0.05mg/kg Dexamethasone for the popliteal nerve block
  Other Names: small dose
  Arms: 0,05mg/kg dexamethasone

SUMMARY:
Effect of Perineural Dexamethasone on the duration of popliteal nerve block for Anesthesia After Pediatric ankle/foot surgery.

DETAILED DESCRIPTION:
This study is proposed to explore the effect of systemic Dexamethasone on the duration of supraclavicular brachial plexus block for analgesia after pediatric ankle surgery.

After foot and ankle surgery, children need good analgesia. Peripheral nerve blocks have provided a safe, effective method to control early postoperative pain when symptoms are most severe.

The safety of local anesthesia is essential in children due to the much lower toxicity threshold of local anesthetics. An effective adjuvant, such as Dexamethasone, could allow for a higher dilution of local anesthetics while maintaining and enhancing their analgesic effect.

There is considerable research where intravenous and perineural dexamethasone use has been compared in adults. However, there is a massive lack of research regarding children.

In this study, investigators compare different doses of perineural Dexamethasone. Groups 2 and 3 have dexamethasone doses of 0.1mg/kg and 0.05mg/kg added to local anesthetic.

The investigator's goal is to find a dexamethasone dose that is as low as possible but simultaneously covers the need for good pain relief and fast recovery postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* children scheduled for hand/wrist surgery
* body weight > 5kg

Exclusion Criteria:

* infection at the site of the regional blockade
* coagulation disorders
* immunodeficiency
* ASA= or >4
* steroid medication in regular use

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2024-02-23 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
first need of opiate | 48 hours
  Time after surgery when the patient needs opiate for the first time

SECONDARY OUTCOMES:
Opioid Consumption | 48 hours
  Total opiate consumption after surgery
Pain score | 4 hours, 8 hours, 12 hours, 16 hours, 18 hours, 24 hours, 28 hours, 32 hours, 36 hours, 40 hours, 44 hours, 48 hours after surgery
  children <3years old FLACC score (Face, Legs, Activity, Cry, Consolability) children >3years old NRS (Numerical Rating Scale)
Blood glucose | 24 and 48 hours after surgery
  Blood glucose every 24 hours during hospitalization
NLR | 24 and 48 hours after surgery
  Neutrophil-to-lymphocyte ratio
PLR | 24 and 48 hours after surgery
  Platelet-to-lymphocyte ratio
Mobilisation | 4 hours, 8 hours, 12 hours, 16 hours, 18 hours, 24 hours, 28 hours, 32 hours, 36 hours, 40 hours, 44 hours, 48 hours after surgery
  Toe movement every 4 hours

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Kotwicki, Prof.dr hab., Study Director — Poznan University of Medical Sciences
Locations (1):
- Poznan University of Medical Sciences, Poznan, Poznań, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reysner M, Reysner T, Janusz P, Kowalski G, Shadi M, Daroszewski P, Wieczorowska-Tobis K, Kotwicki T. Dexamethasone as a perineural adjuvant to a ropivacaine popliteal sciatic nerve block for pediatric foot surgery: a randomized, double-blind, placebo-controlled trial. Reg Anesth Pain Med. 2025 Dec 5;50(12):970-976. doi: 10.1136/rapm-2024-105694. PMID 39209730